CLINICAL TRIAL: NCT01832389
Title: Does a PiCCO-controlled Advanced Haemodynamic Monitoring Improve the Outcome After Aneurysmal Subarachnoid Haemorrhage?
Brief Title: Goal Directed Therapy After Aneurysmal Subarachnoid Haemorrhage
Acronym: PiSAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PiSAH
Record Dates: First submitted 2012-10-29; First posted 2013-04-16 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Aneurysmal Subarachnoid Haemorrhage; SAH
Keywords: Subarachnoid Haemorrhage (SAH); vasospasm; delayed cerebral ischaemia (DCI); goal directed therapy (GDT); Pulse Contour Cardiac Output (PiCCO)
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group P (Active Comparator): PiCCO-controlled group
  Interventions: Device: PiCCO
- Group C (No Intervention): control group

INTERVENTIONS:
Device: PiCCO
  Arms: Group P

SUMMARY:
The objective of this study is to determine whether a goal-directed therapy can reduce the incidence of delayed cerebral ischaemia after aneurysmal subarachnoid haemorrhage.

DETAILED DESCRIPTION:
The aneurysmal subarachnoid haemorrhage (SAH) is a frequent and dangerous worldwide cause for stroke. A typical complication presents delayed cerebral ischemia as a consequence of cerebral vasospasms, which occurs in 46% of the cases. The Triple-H-therapy (Hypervolaemia, Hypertension and Haemodilution) was favoured to prevent ischaemic complications after vasospasm for a long time. However recently, the focus is mainly on hypertension, and it is recommended to maintain normovolaemia. The debate how to assure normovolaemia is still on going, therefore, this study was designed to examine whether a PiCCO-controlled haemodynamic monitoring and a goal-directed therapy can reduce the incidence of delayed cerebral ischaemia after SAH.

The present study is a prospective randomized controlled clinical study. Patients older than 18 years with an aneurysmal SAH will be enrolled. They will be divided into two groups: a control group "C" and a PiCCO group "P". Both groups will be treated according to the current guidelines. In addition, in group P the volume and catecholamine therapy will be controlled by means of PiCCO-controlled monitoring and an algorithm.

The primary end point is the number of occurred delayed cerebral ischaemia per patient. Secondary end points are neurological, pulmonary, cardiovascular, renal, and hepatic complications as well as electrolyte and serum glucose disturbance, sepsis, and mortality, length of hospital and intensive care unit stay and the amount of volume and catecholamines administered.

All participants are to be contacted three months after discharge, and their health status is to be determined by using the GOS (Glasgow Outcome Scale).

ELIGIBILITY:
Inclusion Criteria:

* aneurysmal Subarachnoid Haemorrhage (SAH)
* Age ≥ 18 years

Exclusion Criteria:

* traumatic SAH
* congestive heart failure
* severe diseases of aorta or aortic valve
* pregnancy
* calcium antagonist intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
number of occurred delayed cerebral ischaemia (DCI) per patient | 14 days
  a 2 point increase in the score of the NIHSS-scale lasting for at least 8 hours or a ≥ 2-point decrease in the Glasgow Coma Scale (GCS) lasting for at least 8 hours (as signs of a new focal neurological deficit); and/or radiologic signs of cerebral infarction in presence of vasospasm. other causes of neurological aggravation (e.g. hydrocephalus, re-bleeding etc) had to be excluded.

SECONDARY OUTCOMES:
pulmonary and cardiovascular complications | 3 months
neurological complications | 3 months
renal and hepatic complications | 3 months
electrolyte and serum glucose disturbance | 3 months
sepsis, and mortality | 3 months
length of hospital and intensive care unit stay | 3 months
amount of volume and catecholamines administered | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München; Aida Anetsberger, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, München, Germany

REFERENCES:
- [Background] Suarez JI, Tarr RW, Selman WR. Aneurysmal subarachnoid hemorrhage. N Engl J Med. 2006 Jan 26;354(4):387-96. doi: 10.1056/NEJMra052732. No abstract available. PMID 16436770
- [Derived] Althouse AD, Jain SK, Shalaby A, Singh M, Weiss R, Myaskovsky L, Al-Khatib SM, Saba S. Feasibility of a Randomized Clinical Trial of Cardiac Resynchronization Therapy With or Without an Implantable Defibrillator in Older Patients. Circ Arrhythm Electrophysiol. 2022 Apr;15(4):e010795. doi: 10.1161/CIRCEP.121.010795. Epub 2022 Mar 31. No abstract available. PMID 35357219
- [Derived] Anetsberger A, Gempt J, Blobner M, Ringel F, Bogdanski R, Heim M, Schneider G, Meyer B, Schmid S, Ryang YM, Wostrack M, Schneider J, Martin J, Ehrhardt M, Jungwirth B. Impact of Goal-Directed Therapy on Delayed Ischemia After Aneurysmal Subarachnoid Hemorrhage: Randomized Controlled Trial. Stroke. 2020 Aug;51(8):2287-2296. doi: 10.1161/STROKEAHA.120.029279. Epub 2020 Jul 9. PMID 32640940